CLINICAL TRIAL: NCT04909398
Title: New Methods of Dynamic Pupillometrics in Subjects With Visual and Color Vision Pathologies for the Detection, Functional Diagnosis and Follow-up of These Pathologies
Brief Title: Pupil Dynamics and Color Vision for the Detection of Eye Diseases
Acronym: PupDyn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Streetlab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P17-05
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Retinitis Pigmentosa; Leber's Hereditary Optic Neuropathy; Stargardt Disease
MeSH Terms: conditions — Retinitis Pigmentosa; Optic Atrophy, Hereditary, Leber; Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic pupillometry sessions (Experimental): It is planned to include 60 participants divided into different groups:
  * 15 healthy subjects, called controls.
  * 15 patients with retinitis pigmentosa.
  * 15 patients with Leber's hereditary optic neuropathy.
  * 15 patients with Stargardt's disease.
  Interventions: Behavioral: Dynamic pupillometry sessions

INTERVENTIONS:
Behavioral: Dynamic pupillometry sessions — The evaluation protocol will include the following steps:
  * Installation of the subject, adaptation of the chin rest for the best comfort of the participant
  * Calibration of the oculometer consisting of ocular fixation of 9 fixation points distributed on the stimulation screen
  * Final validation of the eligibility of the subject in the study according to the success or not of the calibration.

SUMMARY:
The development of new oculometry techniques allows fine and dynamic measurements of pupillary diameter and use in routine clinical practice.

The preliminary results obtained with innovative devices on healthy sjuets make it possible to envisage a clinical study on a population of patients suffering from retinal pathologies.

This is a "proof of concept" study, which, if the expected results are confirmed, will make it possible to consider a study on a larger population, as well as the industrial development of a commercial device.

DETAILED DESCRIPTION:
This is a single-head study that will take place at the National Ophthalmology Hospital Center (CHNO) and the Vision Institute (Streetlab) and the total duration of the study is 24 months .

It is planned to include 60 participants divided into different groups:

* 15 healthy subjects, called controls.
* 15 patients with retinitis pigmentosa.
* 15 patients with Leber's hereditary optic neuropathy.
* 15 patients with Stargardt's disease.

Patients will be pre-selected on files at the CHNO clinical investigation center based on the visual assessment carried out on the day of their arrival, the doctor may suggest that they participate in the study if the inclusion criteria are respected.

The control subjects will be recruited thanks to the database of the Vision Institute at Streetlab.

ELIGIBILITY:
Inclusion Criteria:

- Patients with an understanding of the French language to ensure a perfect understanding of the instructions during evaluations and documents relating to their involvement in the study.

Visually impaired volunteers:

Patients must have one of three conditions: Retinitis Pigmentosa, Stargardt disease, Leber optic neuropathy.

Healthy volunteers:

* Visual acuity of both corrected eyes (glasses) should be higher or equal 8/10th and a normal visual field.
* Patients should not wear contact lenses (which may interfere with the recording of the pupil and eye movements)

Exclusion Criteria:

* Pregnant or lactating women will not be able to participate in this research.
* Participants should not be unable to personally consent.
* Subjects should not participate in another clinical trial that may interfere with this research.
* Inability to personally consent.
* Subjects should not present with degenerative diseases or any other disease that could interfere with the evaluations planned during this study.
* The subject follows a drug treatment which can cause visual disturbances, changes in pupillary kinetics or cognitive disturbances.

Secondary exclusion criteria (at the end of the inclusion visit):

* Visually impaired subjects and controls for which calibration is not feasible.
* Patients and control subjects having difficulty maintaining visual fixation.
* Patients and subjects wearing corrective lenses making it impossible to record oculomotor activity with an infrared camera oculometer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Dynamic pupillometry sessions pupillary reflex measurement | Week 1
  Measurement of the right eye / left eye and binocular monocular pupillary reflex: pupillary response measured for 5 seconds with 3 levels of screen luminance, each stimulation will be separated from the next by a delay of 5 seconds
RAPD measurement | Week 1
  Alternate stimulation of the right and left eye: 10 repetitions, each corresponding to the stimulation of one eye for one second.
Endogenous pupillary oscillation measurement | Week 1
  Pupil oscillation frequency, for each eye and in binocular: during this test the participants observe the stimulation screen (central fixation point) for 45 seconds during which the lumnance of the screen is calculated to be proportional to the size of the pupil
  in real time.
Measurement of pupillary activity by frequency marking | Week 1
  This test consists of the simultaneous presentation of 5 areas of the screen, each of which is luminance modulated at a specific frequency.
Pupillary measurement of color vision | Week 1
  In this test, 2 background colors alternate at low frequency over time.
  The physical luminance of one color is fixed while the other is adaptively changed during a test to reduce pupillary response.

CONTACTS AND LOCATIONS:
Overall Officials: Saddek MOHAND-SAID, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National D'Ophtalùmologie des Quinze-Vingts, Paris, France